CLINICAL TRIAL: NCT04181580
Title: Explorative, Monocentric, Feasibility Study Focusing on Fit of Innovative, Made-to-measure Compression Garments in Healthy Subjects
Brief Title: Feasibility Study Focusing on Fit of Made-to-measure Compression Garments in Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BSN Medical GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BSN-C2593
Record Dates: First submitted 2019-11-26; First posted 2019-11-29 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Product Use Issue

STUDY DESIGN:
Intervention Model Description: Healthy subjects will test made-to-measure compression garments. No comparator group due to exploartive design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fit test of made-to-measure garments (Other): Healthy subjects will test maximum 2 compression garments out of 6 garments under investigation
  Interventions: Device: Made-to-measure compression garment

INTERVENTIONS:
Device: Made-to-measure compression garment — Made-to-measure compression garment

SUMMARY:
Fit of made-to-measure compression garments in healthy subjects will be tested on one day, simulating daily activities.

DETAILED DESCRIPTION:
Lower and upper extremities of 36 health subjects will be measured be trained experts to collect measures for made-to-measure compression garments.

Fit of made-to-measure compression garments, which are not on the market yet, among healthy subjects will be tested on one day, simulating daily activities. Fit will be assessed directly after donning and after a wearing period of maximum 7 hours at the study site by trained experts. Healthy subjects will give back study products at the end of the wearing period. AEs will be documented throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Men, women or diverse
* Full legal competence
* Age between 18 and 70 years
* Capability to understand the subject information and to provide conscious informed consent
* All female or diverse subjects of childbearing potential must either be surgically sterile (hysterectomy or tubal ligation) or agree to use a reliable method of contraception with a Pearl-Index of less than 1% per year when used consistently and correctly such as implants, injectables, combined oral contraceptives, some intra uterine devices (IUDs), sexual abstinence or vasectomized partner for at least 4 weeks
* Willingness to conduct a urine pregnancy test for all females or potentially childbearing diverse subjects
* Capability and willingness to follow protocol requirements
* Signed informed consent for study participation and data protection regulations
* Body mass index (BMI) >23 kg/m² and ≤ 40 kg/m²

Exclusion Criteria:

* Circumference of the largest circumference of the upper leg >80 cm (measured in the upright position)
* Shape distortions
* Diagnosed lymphedema of the upper and/or lower extremities
* Diagnosed lipedema of upper and/or lower extremities
* Diagnosed indication for therapy with flat-knitted compression garments
* Alcohol abuse as reported by subject and/ or suspected by investigator
* Drug abuse as reported by subject and/ or suspected by investigator
* Allergy or sensitivity to one or more components of the investigational devices, as far as reported by the subject
* Circumference of the largest circumference of the upper leg >80 cm (measured in the upright position)
* Shape distortions
* Diagnosed lymphedema of the upper and/or lower extremities
* Diagnosed lipedema of upper and/or lower extremities
* Diagnosed indication for therapy with flat-knitted compression garments
* Alcohol abuse as reported by subject and/ or suspected by investigator
* Drug abuse as reported by subject and/ or suspected by investigator
* Allergy or sensitivity to one or more components of the investigational devices, as far as reported by the subject
* Pregnancy or breastfeeding
* Diagnosed peripheral arterial disease
* Presence of untreated phlebitis, or septic phlebitis
* Diagnosed progressed arterial insufficiency including ischemia
* Diagnosed congestive heart failure
* Diagnosed clinically relevant hypertension
* Diagnosed renal insufficiency or kidney failure
* Presence of Untreated or progressing skin infection
* Presence of large coagulum in the leg vein
* Presence of phlegmasia coerulea dolens
* Diagnosed Raynaud's disease
* Diagnosed gonarthrosis
* Diagnosed ankle arthrosis
* Diagnosed rheumatoid arthritis
* Presence of Exuding dermatoses
* Presence of gangrene
* Diagnosed malign lymphedema
* Diagnosed psoriasis
* Diagnosed diabetes mellitus
* Diagnosed complex regional pain syndrome (CRPS; Sudeck atrophy)
* Diagnosed polyneuropathy
* Diagnosed severe impaired skin sensitivity und impaired sensitivity of the extremities, including all sensory malfunctions and diagnosed impaired pain sensitivity
* Objections of the investigator to the subject's participation in the trial due to medical reasons or any other reason for which the subject should not participate in the opinion of the investigator
* Participation in any clinical investigation with systemic and/or pharmaceutical substances within the last 4 weeks and/or in parallel
* Sponsors, manufacturers or CRO staff

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-11-28 (Actual); Primary Completion 2019-12-13 (Actual); Study Completion 2019-12-13 (Actual)

PRIMARY OUTCOMES:
Evaluation of the fit of the investigational device | One day
  Evaluation of the fit of the investigational medical device at the end of a wearing period of approximately 4 - 7 hours by predefined criteria, to be worn by healthy subjects once.

CONTACTS AND LOCATIONS:
Overall Officials: Uwe Kröncke, Principal Investigator — Bioskin GmbH
Locations (1):
- bioskin GmbH, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared. Data are needed for confidential medical device development.